CLINICAL TRIAL: NCT03957226
Title: An Osseoanchored Percutaneous Prosthesis Study Evaluating Stable Neural Signal Transmission in Subjects With Transhumeral Amputations
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was not sufficiently funded. No enrollment took place.
Sponsor: University of Michigan (Other)
Collaborators: University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Paul Cederna, Robert Oneal Professor of Plastic Surgery, Chief of the Section of Plastic Surgery, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: HUM00146699
Record Dates: First submitted 2019-05-02; First posted 2019-05-21 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-10

CONDITIONS: Amputation Neuroma; Amputation; Prosthesis User

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Trasnhumeral e-OPRA Implant (Experimental): This arm includes patients with transhumeral amputation that will receive the e-OPRA implant system.
  Interventions: Device: e-OPRA (electronic-Osseoanchored Prosthese for the Rehabilitation of Amputees)

INTERVENTIONS:
Device: e-OPRA (electronic-Osseoanchored Prosthese for the Rehabilitation of Amputees) — The e-OPRA is an implant system that provides an alternative to traditional socket prostheses by establishing a direct, load-bearing link between the patient's skeleton and a prosthesis for transhumeral amputees. The anchorage element of the system is implanted directly into the bone while the electrodes that provide control signals for the prosthesis are implanted into muscle grafts on the transhumeral amputation.

SUMMARY:
This early feasibility study proposes to evaluate use of the electronic-Osseoanchored Prostheses for the Rehabilitation of Amputees (e-OPRA) device, a transhumeral implant system for direct skeletal anchorage of amputation prostheses, with a test prosthesis. The e-OPRA System is being investigated to better understand the ability to improve the functionality of the prosthesis and enhance the sense of embodiment of the prosthesis itself. This will be a 10 subject Early Feasibility Study in which the primary objective is to capture preliminary safety and effectiveness information on the implanted e-OPRA system. With the addition of electrodes to the muscle segments, this biological interface allows for both the extraction of fine motor control signals from the nerve fascicles and the generation of sensory percepts via electrical stimulation of the muscles. In addition, electrodes placed on muscles within the residuum with native vascularization and innervation also allow the extraction of critical motor control signals and the generation of sensory feedback through muscle stimulation. The electrical activity recorded from these muscle segments (called electromyography or EMG) is specific to certain movements and can be used to determine precisely how a person wants to move their arm and hand. Use of the e-OPRA device with the well-documented neuro-electronic capabilities of EMG control systems provides an alternative to traditional socket prostheses by establishing a direct, loadbearing link between the patient's skeleton and prosthesis.

ELIGIBILITY:
Inclusion Criteria:

* Male or female age 22-65 at the time of surgery.
* The patient must have one of the following medical conditions:

  * A condition requiring performance of a unilateral transhumeral amputation;
  * An existing transhumeral OPRA device implanted under IDE G150155;
  * An existing unilateral transhumeral amputation; or
  * An existing unilateral transhumeral amputation with previous nerve reinnervation surgery.
* The patient must have a residual humerus of greater than or equal to 10 cm.
* The patient must have a cortical thickness of at least 1.5 mm.
* The patient must have at least a portion of biceps and triceps muscles present.
* The subject must have undergone consultation with at least two upper extremity surgical specialists to ensure they have exhausted all limb salvage options prior to undergoing amputation.
* The patient must have adequate bone stock to support the implanted device.
* In the opinion of the Investigators, normal cognitive function and absence of any physical limitations, addictive diseases or underlying medical conditions that may preclude patient from being a good surgical and/or study candidate.
* Willingness, ability and commitment to participate in baseline and follow-up evaluations for the full length of the study including the prescribed rehabilitation program.
* Written informed consent to participate in the study provided by the patient or legal representative.

Exclusion Criteria:

* Women who are pregnant, lactating, or planning a pregnancy during the first twelve (12) months of the post-surgical follow-up.
* Arthrosis of the ipsilateral glenohumeral joint by radiographs.
* Subjects who have not been completely abstinent from tobacco use for at least 6 weeks preoperatively.
* Active or dormant infection.
* Evidence of or a documented history of severe peripheral vascular disease, diabetes mellitus (type I or type II), skin diseases, neuropathy, neuropathic disease, severe phantom pain, or osteoporosis, such that, in the opinion of the Investigator, the subject will not be a good study candidate.
* History of systemically administered corticosteroids, immunosuppressive therapy, or chemotherapeutic drugs within six (6) months of implant surgery.
* Severe medical co-morbidity, atypical skeletal anatomy, or poor general physical/mental health that, in the opinion of the Investigator, will not allow the subject to be a good study candidate (i.e., other disease processes, other indwelling electronic implants, mental incapacity, substance abuse, shortened life expectancy, and vulnerable patient population).
* Current involvement in another clinical study where that participation may conflict or interfere with the treatment, follow-up or results of this clinical study.

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-01-30 (Estimated); Primary Completion 2022-06-23 (Actual); Study Completion 2022-06-23 (Actual)

PRIMARY OUTCOMES:
Change in Electrical signal quality between implanted electrodes and test prosthesis | Baseline, 24 months
  Efficacy will be evaluated by signal-to-noise ratio during maximum voluntary contraction of at least two independent myoelectric signals.
Adverse Events | Baseline
  Safety will be evaluated by assessing the adverse event type, incidence, timing, severity, treatment, outcome, and relationship to the device.
Adverse Events | 3 Months Post-Op
  Safety will be evaluated by assessing the adverse event type, incidence, timing, severity, treatment, outcome, and relationship to the device.
Adverse Events | 6 Months Post-Op
  Safety will be evaluated by assessing the adverse event type, incidence, timing, severity, treatment, outcome, and relationship to the device.
Adverse Events | 9 Months Post-Op
  Safety will be evaluated by assessing the adverse event type, incidence, timing, severity, treatment, outcome, and relationship to the device.
Adverse Events | 12 Months Post-Op
  Safety will be evaluated by assessing the adverse event type, incidence, timing, severity, treatment, outcome, and relationship to the device.
Adverse Events | 15 Months Post-Op
  Safety will be evaluated by assessing the adverse event type, incidence, timing, severity, treatment, outcome, and relationship to the device.
Adverse Events | 18 Months Post-Op
  Safety will be evaluated by assessing the adverse event type, incidence, timing, severity, treatment, outcome, and relationship to the device.
Adverse Events | 21 Months Post-Op
  Safety will be evaluated by assessing the adverse event type, incidence, timing, severity, treatment, outcome, and relationship to the device.
Adverse Events | 24 Months Post-Op
  Safety will be evaluated by assessing the adverse event type, incidence, timing, severity, treatment, outcome, and relationship to the device.

SECONDARY OUTCOMES:
Number of Subjects with 2 or more Degrees of Freedom | Baseline, 24 months
  The number of subjects achieving 2 or more degrees of freedom summarized using frequency and percentage
Change in Pain Level as measured by SF-36 | Baseline, 24 months
  Change in Pain Level as measured by SF-36 survey Pain will be assessed using the SF-36 survey instrument, to be filled out by the participant before and after each surgical procedure performed and at a minimum of once per month while electrodes remain implanted. Scores range from 0 - 100 Lower scores = more disability, higher scores = less disability.
Change in Pain Level as measured by LANSS surveys | Baseline, 24 months
  Change in Pain Level as measured by LANSS survey Pain will be assessed using the LANSS survey instrument, to be filled out by the participant before and after each surgical procedure performed and at a minimum of once per month while electrodes remain implanted. A score greater than 12 (From 0 to 15) indicates neuropathic pain.
Change in prosthetic functionality and performance as measured by the SHAP (Southhampton Hand Assessment Procedure) | Baseline, 24 months
  Measured by the participant performing the SHAP at each experimental visit. A higher score indicates increased upper limb functionality.
Change in prosthetic functionality and performance as measured by the AM-ULA (Activities Measure for Upper Limb Amputees) | Baseline, 24 months
  Measured by the participant performing the AM-ULA at each experimental visit. A higher score indicates increased upper limb functionality.
Change in prosthetic functionality and performance as measured by the UEFT (Upper Extremity Function Test) | Baseline, 24 months
  Measured by the participant performing the UEFT at each experimental visit. A higher score indicates increased upper limb functionality.
Change in Pain Level as measured by PROMIS (Patient Reported Outcomes Measurement Information System) Questionnaire | Baseline, 24 months
  Change in Pain Level as measured by LANSS survey Pain will be assessed using the LANSS survey instrument, to be filled out by the participant before surgery and at each experimental visit. The Numeric Rating Scale measures (adult, pediatric, parent proxy) each consist of a single item rating pain on average over the past 7 days from 0 (no pain) to 10 (worst pain you can think of). The items are not calibrated and do not produce a T-score. Instead, raw response scores (0 to 10) should be used for analyses.
Change in prosthetic functionality as measured by the DASH Questionnaire | Baseline, 24 months
  Measured by the participant filling out the DASH questionnaire before surgery and at each experimental visit every 3 months. A score closer to 1 indicates higher functionality. The DASH Outcome Measure is scored in two components: the disability/symptom section (30 items, scored 1-5) and the optional high performance Sport/Music or Work section (4 items, scored 1-5). The raw is transformed to a zero-to-100 scale, with an average score closer to 100 meaning higher disability (unable to perform tasks).
Change in Pain Level as measured by DVPRS (Defense and Veterans Pain Rating Scale) | Baseline, 24 months
  Measured by the participant assigning a number 1-10 of their pain while viewing the DVPRS. A score close to of 0 indicates zero pain, and a score of 10 indicates maximum pain as bad is it can be.
Change in Quality of Life as measured by the EQ-5D-5L Questionnaire | Baseline, 24 months
  Measured by the participant filling out the EQ-5D-5L before surgery and at each experimental visit every 3 months. Each question is scored from 1-5, with 5 having the most difficulty in that area.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Cederna, MD, Principal Investigator — University of Michigan, Section of Plastic Surgery
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States